CLINICAL TRIAL: NCT01001351
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study of a Single Dose of PRT-201 Administered Immediately After Arteriovenous Graft Creation in Patients With Chronic Kidney Disease
Brief Title: A Study of PRT-201 Administered After Arteriovenous Graft (AVG) Creation in Patients With Chronic Kidney Disease
Acronym: PRT-201-102
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Proteon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PRT-201-102
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Arteriovenous Grafts (AVG); Hemodialysis; Vascular Access; Dialysis; Graft; Access; vonapanitase; kidney; renal
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — cholesterol-binding protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PRT-201 (Experimental)
  Interventions: Drug: PRT-201

INTERVENTIONS:
Drug: PRT-201 — Applied topically during surgery.
  Arms: PRT-201
Drug: Placebo — Applied topically during surgery
  Arms: Placebo

SUMMARY:
PRT-201 is a recombinant human type-I pancreatic elastase intended for local, long-lasting dilation of the AVG venous anastomosis and outflow vein. The goal of the treatment is to improve primary patency and long-term survival of AVGs and thereby provide patients with chronic kidney disease (CKD) a reliable and durable vascular access site for hemodialysis. Recent data indicate that up to three quarters of patients have loss of graft patency at one year, indicating a substantial need for new therapies. This clinical trial will explore the safety and dilatory effect of topically administered PRT-201 on the outflow vein of a newly placed upper extremity AVG.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 years.
2. Chronic kidney disease with anticipated start of hemodialysis within 3 months or current hemodialysis dependence.
3. Planned creation of a new upper extremity AVG or "jump" graft

Exclusion Criteria:

1. Patients for whom this is the only potential site for an upper extremity vascular access.
2. Creation of a new AVG or "jump" graft in an upper extremity previously treated with an investigational gene or cell based therapy, or locally with an investigational pharmacological agent.
3. On physical examination or by other means, suspected proximal vein stenosis, occlusion, lack of continuity with the subclavian vein, central venous stenosis or central venous occlusion.
4. History or presence of an arterial aneurysm.
5. Previous treatment with PRT-201.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2009-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To assess the safety of a single topical dose of PRT-201. | Day of AVG creation and 4 weeks After surgery.

SECONDARY OUTCOMES:
Primary graft patency | 3, 6, 9 and 12 months after AVG creation.
Secondary graft patency. | 3, 6, 9 and 12 months after AVG creation.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Wong, MD, PhD, Study Director — Proteon Therapeutics, Inc
Locations (16):
- United States (16):
  - Ladenheim Dialysis Access Center, Fresno, California
  - California Institute of Renal Research, San Diego, California
  - Washington Hospital/Medstar Research, Washington D.C., District of Columbia
  - Indiana/Ohio Heart, Fort Wayne, Indiana
  - Indiana University/Purdue University, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Vascular Specialty Center, Baton Rouge, Louisiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Greenville Memorial Hospital, Greenville, South Carolina
  - The Methodist Hospital, Houston, Texas
  - Peripheral Vascular Associates, San Antonio, Texas
  - Sentara Vascular Specialists, Norfolk, Virginia

REFERENCES:
- [Result] Dwivedi AJ, Roy-Chaudhury P, Peden EK, Browne BJ, Ladenheim ED, Scavo VA, Gustafson PN, Wong MD, Magill M, Lindow F, Blair AT, Jaff MR, Franano FN, Burke SK. Application of human type I pancreatic elastase (PRT-201) to the venous anastomosis of arteriovenous grafts in patients with chronic kidney disease. J Vasc Access. 2014 Sep-Oct;15(5):376-84. doi: 10.5301/jva.5000235. Epub 2014 May 3. PMID 24811601
- [Derived] Mohamed I, Kamarizan MFA, Da Silva A. Medical adjuvant treatment to increase patency of arteriovenous fistulae and grafts. Cochrane Database Syst Rev. 2021 Jul 23;7(7):CD002786. doi: 10.1002/14651858.CD002786.pub4. PMID 34298589